CLINICAL TRIAL: NCT07338890
Title: Post-Market Clinical Follow-Up Study of the S.M.A.R.T.™ Nitinol Stent System, S.M.A.R.T.™ CONTROL™ Nitinol Stent System and S.M.A.R.T. ™ Flex Vascular Stent System in the Treatment of Iliac and Femoropopliteal Artery Disease (REAL-SMART)
Brief Title: Post-Market Clinical Follow-Up of S.M.A.R.T. Family of Stents in Treating Iliac and Femoropopliteal Artery Disease
Acronym: REAL-SMART
Status: Not yet recruiting | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Collaborators: Rede Optimus Hospitalar SA (Network)
Responsible Party: Sponsor
Other Study IDs: P24-6202
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Superficial Femoral Artery Stenosis; Iliac Artery Stenosis; Popliteal Artery Stenosis
Keywords: Superficial Femoral Artery Stenosis; Iliac Artery Stenosis; Popliteal Artery Stenosis; SMART CONTROL Nitinol Stent System; SMART FLEX Vascular Stent System; SMART Nitinol Stent System; SFA Stenosis; PPA Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (6):
- Subjects with stenotic lesions of the superficial femoral artery (SFA) treated with SMART 120/150.: The Cordis S.M.A.R.T.TM Nitinol Stent System (SMART 120/150) is indicated in enabling treatment in patients with atherosclerotic disease of the superficial femoral artery (SFA).
  Interventions: Device: S.M.A.R.T.™ Nitinol Stent System (SMART 120/150)
- Subjects with stenotic lesions of the proximal popliteal artery (PPA) treated with SMART 120/150.: The Cordis S.M.A.R.T.TM Nitinol Stent System (SMART 120/150) is indicated in enabling treatment in patients with atherosclerotic disease of the proximal popliteal artery (PPA).
  Interventions: Device: S.M.A.R.T.™ Nitinol Stent System (SMART 120/150)
- Subjects with stenotic lesions of the iliac artery treated with SMART CONTROL.: The Cordis S.M.A.R.T.TM CONTROLTM Nitinol Stent System is indicated in enabling treatment in patients with atherosclerotic disease of the iliac artery.
  Interventions: Device: S.M.A.R.T.™ CONTROL ™ Nitinol Stent System
- Subjects with stenotic lesions of the superficial femoral artery (SFA) treated with SMART CONTROL.: The Cordis S.M.A.R.T.TM CONTROLTM Nitinol Stent System is indicated in enabling treatment in patients with atherosclerotic disease of the superficial femoral artery (SFA).
  Interventions: Device: S.M.A.R.T.™ CONTROL ™ Nitinol Stent System
- Subjects with stenotic lesions of the superficial femoral artery (SFA) treated with SMART Flex.: The Cordis S.M.A.R.T.TM Flex Stent is indicated in enabling treatment of patients with symptomatic vascular stenotic and/or occlusive diseases in the superficial femoral artery (SFA).
  Interventions: Device: S.M.A.R.T.™ Flex Vascular Stent System
- Subjects with stenotic lesions of the proximal popliteal artery (PPA) treated with SMART Flex.: The Cordis S.M.A.R.T.TM Flex Stent is indicated in enabling treatment of patients with symptomatic vascular stenotic and/or occlusive diseases in the proximal popliteal artery (PPA).
  Interventions: Device: S.M.A.R.T.™ Flex Vascular Stent System

INTERVENTIONS:
Device: S.M.A.R.T.™ Nitinol Stent System (SMART 120/150) — The Cordis S.M.A.R.T.™ Nitinol Stent System is intended to deliver a self-expanding endovascular stent to the peripheral vasculature via a sheathed delivery system. The stent component imparts an outward radial force on the luminal surface of the vessel wall restoring vascular patency. The S.M.A.R.T. ™ Nitinol Stent System is indicated in enabling treatment in patients with atherosclerotic disease of the superficial femoral artery and proximal popliteal artery.
  Groups: Subjects with stenotic lesions of the proximal popliteal artery (PPA) treated with SMART 120/150.; Subjects with stenotic lesions of the superficial femoral artery (SFA) treated with SMART 120/150.
Device: S.M.A.R.T.™ CONTROL ™ Nitinol Stent System — The Cordis S.M.A.R.T.™ CONTROL™ Nitinol Stent System is intended to deliver a self-expanding endovascular stent to the iliac and/or superficial femoral arteries via a sheathed delivery system. The stent component imparts an outward radial force on the luminal surface of the vessel wall restoring vascular patency. The S.M.A.R.T. ™ CONTROL™ Nitinol Stent System is indicated in enabling treatment in patients with atherosclerotic disease of iliac and/or superficial femoral arteries.
  Groups: Subjects with stenotic lesions of the iliac artery treated with SMART CONTROL.; Subjects with stenotic lesions of the superficial femoral artery (SFA) treated with SMART CONTROL.
Device: S.M.A.R.T.™ Flex Vascular Stent System — The Cordis S.M.A.R.T.™ Flex Stent is a single-use device consisting of an endovascular stent and sheath delivery system, intended to deliver a self-expanding endovascular stent to the superficial femoral artery (SFA). The stent component imparts an outward radial force on the luminal surface of the vessel wall restoring vascular patency. The S.M.A.R.T.™ Flex Stent is indicated in enabling treatment of patients with symptomatic vascular stenotic and/or occlusive diseases in the superficial femoral artery and proximal popliteal artery.
  Groups: Subjects with stenotic lesions of the proximal popliteal artery (PPA) treated with SMART Flex.; Subjects with stenotic lesions of the superficial femoral artery (SFA) treated with SMART Flex.

SUMMARY:
The purpose of this study is to evaluate long-term safety and performance per the intended use of the S.M.A.R.T.™ Nitinol Stent System (SMART 120/150), S.M.A.R.T.™ CONTROL™ Nitinol Stent System (SMART CONTROL) and S.M.A.R.T.™ Flex Vascular Stent System (SMART Flex) in the treatment of iliac and femoropopliteal artery disease.

DETAILED DESCRIPTION:
The REAL-SMART study is a multi-center, non-randomized, observational analysis of retrospective data collected on all subjects treated with SMART 120/150, SMART CONTROL or SMART Flex. The purpose of this study is to evaluate long-term safety and performance per the intended use of the three (3) study devices. Each device constitutes a separate study arm and each arm is further stratified by indication, of which there are two per device. The study is conducted in approximately 20 sites located in approximately three (3) European countries with high volume use of one or more of the study devices. The enrollment and data collection take approximately 6-8 months.

ELIGIBILITY:
Inclusion Criteria: For data mining purposes, the following criteria will apply in determining which subjects to include in the study:

* Subjects treated with SMART 120/150, SMART CONTROL or SMART Flex according to the respective Instructions for Use for treatment in the iliac, superficial femoral and/or proximal popliteal arteries.
* If an EC-approved informed consent waiver is not obtained, then documented informed consent from the subject or legal representative granting permission to share the subject's clinical data It is recommended to include subjects with follow-up data available for a minimum of five (5) years from the date of treatment/procedure or until time of death, whichever came first.

It is recommended to include subjects with follow-up data available for a minimum of five (5) years from the date of treatment/procedure or until time of death, whichever came first. Subjects not included because follow-up information is unavailable will be documented, wherever possible, with respect to demographics and presenting disease state to determine whether they are similar to subjects with follow-up that are enrolled.

Exclusion Criteria: For data mining purposes, the following criteria will apply in determining which subjects to exclude in the study:

* Women who were pregnant or lactating at the time of the procedure.
* Pediatric subjects (<18 years of age) at the time of the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects to be included in this study are those treated with SMART 120/150, SMART CONTROL or SMART Flex, according to the respective Instructions for Use, for stenosis in the iliac, superficial femoral and/or proximal popliteal arteries. Approximately 20 sites located in approximately three (3) European countries with high volume use of one or more of the study products will participate.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Technical success of SMART 120/150 in patients with obstructive SFA disease | At the conclusion of the index procedure
  Technical success, defined as achievement of a final diameter stenosis of less than or equal to (≤) 30% residual stenosis at the conclusion of the index procedure
Major amputation in patients treated with SMART 120/150 for obstructive SFA disease | At 12 months post-index procedure
  Major amputation at 12 months post-index procedure
Technical success of SMART 120/150 in patients with obstructive PPA disease | At the conclusion of the index procedure
  Technical success, defined as achievement of a final diameter stenosis of less than or equal to (≤) 30% residual stenosis at the conclusion of the index procedure
Major amputation in patients treated with SMART 120/150 for obstructive PPA disease | At 12 months post-index procedure
  Major amputation at 12 months post-index procedure
Technical success of SMART CONTROL in patients with obstructive iliac artery disease | At the conclusion of the index procedure
  Technical success, defined as achievement of a final diameter stenosis of less than or equal to (≤) 30% residual stenosis at the conclusion of the index procedure
Major amputation in patients with SMART CONTROL for obstructive iliac artery disease | At 12 months post-index procedure
  Major amputation at 12 months post-index procedure
Technical success of SMART CONTROL in patients with obstructive SFA disease | At the conclusion of the index procedure
  Technical success, defined as achievement of a final diameter stenosis of less than or equal to (≤) 30% residual stenosis at the conclusion of the index procedure
Major amputation in patients treated with SMART CONTROL for obstructive SFA disease | At 12 months post-index procedure
  Major amputation at 12 months post-index procedure
Technical success of SMART Flex in patients with obstructive SFA disease | At the conclusion of the index procedure
  Technical success, defined as achievement of a final diameter stenosis of less than or equal to (≤) 30% residual stenosis at the conclusion of the index procedure
Major amputation in patients treated with SMART Flex for obstructive SFA disease | At 12 months post-index procedure
  Major amputation at 12 months post-index procedure
Technical success of SMART Flex in patients with obstructive PPA disease | At the conclusion of the index procedure
  Technical success, defined as achievement of a final diameter stenosis of less than or equal to (≤) 30% residual stenosis at the conclusion of the index procedure
Major amputation in patients treated with SMART Flex for obstructive PPA disease | At 12 months post-index procedure
  Major amputation at 12 months post-index procedure

SECONDARY OUTCOMES:
Patency at 12 months post-index procedure in patients treated with SMART 120/150 for obstructive SFA disease | At 12 months post-index procedure
  Patency at 12 months post-index procedure, defined as achievement of less than or equal to (≤) 50% diameter stenosis
Patency at 12 months post-index procedure in patients treated with SMART 120/150 for obstructive PPA disease | At 12 months post-index procedure
  Patency at 12 months post-index procedure, defined as achievement of less than or equal to (≤) 50% diameter stenosis
Patency at 12 months post-index procedure in patients treated with SMART CONTROL for obstructive iliac artery disease | At 12 months post-index procedure
  Patency at 12 months post-index procedure, defined as achievement of less than or equal to (≤) 50% diameter stenosis
Patency at 12 months post-index procedure in patients treated with SMART CONTROL for obstructive SFA disease | At 12 months post-index procedure
  Patency at 12 months post-index procedure, defined as achievement of less than or equal to (≤) 50% diameter stenosis
Patency at 12 months post-index procedure in patients treated with SMART Flex for obstructive SFA disease | At 12 months post-index procedure
  Patency at 12 months post-index procedure, defined as achievement of less than or equal to (≤) 50% diameter stenosis
Patency at 12 months post-index procedure in patients treated with SMART Flex for obstructive PPA disease | At 12 months post-index procedure
  Patency at 12 months post-index procedure, defined as achievement of less than or equal to (≤) 50% diameter stenosis
Target lesion restenosis in patients treated with SMART 120/150 for obstructive SFA disease | At 12 months post-index procedure
  Target lesion restenosis, defined as greater than (>) 50% diameter stenosis at 12 months post-index procedure
Target lesion restenosis in patients treated with SMART 120/150 for obstructive PPA disease | At 12 months post-index procedure
  Target lesion restenosis, defined as greater than (>) 50% diameter stenosis at 12 months post-index procedure
Target lesion restenosis in patients treated with SMART CONTROL for obstructive iliac artery disease | At 12 months post-index procedure
  Target lesion restenosis, defined as greater than (>) 50% diameter stenosis at 12 months post-index procedure
Target lesion restenosis in patients treated with SMART CONTROL for obstructive SFA disease | At 12 months post-index procedure
  Target lesion restenosis, defined as greater than (>) 50% diameter stenosis at 12 months post-index procedure
Target lesion restenosis in patients treated with SMART Flex for obstructive SFA disease | At 12 months post-index procedure
  Target lesion restenosis, defined as greater than (>) 50% diameter stenosis at 12 months post-index procedure
Target lesion restenosis in patients treated with SMART Flex for obstructive PPA disease | At 12 months post-index procedure
  Target lesion restenosis, defined as greater than (>) 50% diameter stenosis at 12 months post-index procedure
Procedural success in patients treated with SMART 120/150 for obstructive SFA disease | At the conclusion of the index procedure
  Procedural success, defined as successful stent deployment without occurrence of any procedural complications
Procedural success in patients treated with SMART 120/150 for obstructive PPA disease | At the conclusion of the index procedure
  Procedural success, defined as successful stent deployment without occurrence of any procedural complications
Procedural success in patients treated with SMART CONTROL for obstructive iliac artery disease | At the conclusion of the index procedure
  Procedural success, defined as successful stent deployment without occurrence of any procedural complications
Procedural success in patients treated with SMART CONTROL for obstructive SFA disease | At the conclusion of the index procedure
  Procedural success, defined as successful stent deployment without occurrence of any procedural complications
Procedural success in patients treated with SMART Flex for obstructive SFA disease | At the conclusion of the index procedure
  Procedural success, defined as successful stent deployment without occurrence of any procedural complications
Procedural success in patients treated with SMART Flex for obstructive PPA disease | At the conclusion of the index procedure
  Procedural success, defined as successful stent deployment without occurrence of any procedural complications
Target Lesion Revascularization in patients treated with SMART 120/150 for obstructive SFA disease | Through 12 months post-index procedure
  Target Lesion Revascularization through 12 months post-index procedure
Target Lesion Revascularization in patients treated with SMART 120/150 for obstructive PPA disease | Through 12 months post-index procedure
  Target Lesion Revascularization through 12 months post-index procedure
Target Lesion Revascularization in patients treated with SMART CONTROL for obstructive iliac artery disease | Through 12 months post-index procedure
  Target Lesion Revascularization through 12 months post-index procedure
Target Lesion Revascularization in patients treated with SMART CONTROL for obstructive SFA disease | Through 12 months post-index procedure
  Target Lesion Revascularization through 12 months post-index procedure
Target Lesion Revascularization in patients treated with SMART Flex for obstructive SFA disease | Through 12 months post-index procedure
  Target Lesion Revascularization through 12 months post-index procedure
Target Lesion Revascularization in patients treated with SMART Flex for obstructive PPA disease | Through 12 months post-index procedure
  Target Lesion Revascularization through 12 months post-index procedure
All-Cause Mortality through 30 days post-index procedure in patients treated with SMART 120/150 for obstructive SFA disease | Through 30 days post-index procedure
  All-Cause Mortality through 30 days post-index procedure
All-Cause Mortality through 30 days post-index procedure in patients treated with SMART 120/150 for obstructive PPA disease | Through 30 days post-index procedure
  All-Cause Mortality through 30 days post-index procedure
All-Cause Mortality through 30 days post-index procedure in patients treated with SMART CONTROL for obstructive iliac artery disease | Through 30 days post-index procedure
  All-Cause Mortality through 30 days post-index procedure
All-Cause Mortality through 30 days post-index procedure in patients treated with SMART CONTROL for obstructive SFA disease | Through 30 days post-index procedure
  All-Cause Mortality through 30 days post-index procedure
All-Cause Mortality through 30 days post-index procedure in patients treated with SMART Flex for obstructive SFA disease | Through 30 days post-index procedure
  All-Cause Mortality through 30 days post-index procedure
All-Cause Mortality through 30 days post-index procedure in patients treated with SMART Flex for obstructive PPA disease | Through 30 days post-index procedure
  All-Cause Mortality through 30 days post-index procedure
Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure in patients treated with SMART 120/150 for obstructive SFA disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure
Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure in patients treated with SMART 120/150 for obstructive PPA disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure
Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure in patients treated with SMART CONTROL for obstructive iliac artery disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure
Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure in patients treated with SMART CONTROL for obstructive SFA disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure
Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure in patients treated with SMART Flex for obstructive SFA disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure
Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure in patients treated with SMART Flex for obstructive PPA disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse events (SAE) through 36 months (3 years) post-index procedure
Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure in patients treated with SMART 120/150 for obstructive SFA disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure
Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure in patients treated with SMART 120/150 for obstructive PPA disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure
Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure in patients treated with SMART CONTROL for obstructive iliac artery disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure
Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure in patients treated with SMART CONTROL for obstructive SFA disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure
Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure in patients treated with SMART Flex for obstructive SFA disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure
Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure in patients treated with SMART Flex for obstructive PPA disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse events (SAE) through 60 months (5 years) post-index procedure
Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure in patients treated with SMART 120/150 for obstructive SFA disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure
Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure in patients treated with SMART 120/150 for obstructive PPA disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure
Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure in patients treated with SMART CONTROL for obstructive iliac artery disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure
Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure in patients treated with SMART CONTROL for obstructive SFA disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure
Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure in patients treated with SMART Flex for obstructive SFA disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure
Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure in patients treated with SMART Flex for obstructive PPA disease | Through 36 months (3 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 36 months (3 years) post-index procedure
Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure in patients treated with SMART 120/150 for obstructive SFA disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure
Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure in patients treated with SMART 120/150 for obstructive PPA disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure
Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure in patients treated with SMART CONTROL for obstructive iliac artery disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure
Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure in patients treated with SMART CONTROL for obstructive SFA disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure
Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure in patients treated with SMART Flex for obstructive SFA disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure
Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure in patients treated with SMART Flex for obstructive PPA disease | Through 60 months (5 years) post-index procedure
  Rate of serious adverse device effects (SADE) through 60 months (5 years) post-index procedure
Rate of stent fractures by type at 6 months post-index procedure in patients treated with SMART 120/150 for obstructive SFA disease | At 6 months post-index procedure
  Rate of stent fractures at 6 months post-index procedure
Rate of stent fractures by type at 6 months post-index procedure in patients treated with SMART 120/150 for obstructive PPA disease | At 6 months post-index procedure
  Rate of stent fractures at 6 months post-index procedure
Rate of stent fractures by type at 6 months post-index procedure in patients treated with SMART CONTROL for obstructive iliac artery disease | At 6 months post-index procedure
  Rate of stent fractures at 6 months post-index procedure
Rate of stent fractures by type at 6 months post-index procedure in patients treated with SMART CONTROL for obstructive SFA disease | At 6 months post-index procedure
  Rate of stent fractures at 6 months post-index procedure
Rate of stent fractures at 6 months by type post-index procedure in patients treated with SMART Flex for obstructive SFA disease | At 6 months post-index procedure
  Rate of stent fractures at 6 months post-index procedure
Rate of stent fractures at 6 months by type post-index procedure in patients treated with SMART Flex for obstructive PPA disease | At 6 months post-index procedure
  Rate of stent fractures at 6 months post-index procedure
Rate of stent fractures at 12 months by type post-index procedure in patients treated with SMART 120/150 for obstructive SFA disease | At 12 months post-index procedure
  Rate of stent fractures at 12 months post-index procedure
Rate of stent fractures at 12 months by type post-index procedure in patients treated with SMART 120/150 for obstructive PPA disease | At 12 months post-index procedure
  Rate of stent fractures at 12 months post-index procedure
Rate of stent fractures at 12 months by type post-index procedure in patients treated with SMART CONTROL for obstructive iliac artery disease | At 12 months post-index procedure
  Rate of stent fractures at 12 months post-index procedure
Rate of stent fractures at 12 months by type post-index procedure in patients treated with SMART CONTROL for obstructive SFA disease | At 12 months post-index procedure
  Rate of stent fractures at 12 months post-index procedure
Rate of stent fractures at 12 months by type post-index procedure in patients treated with SMART Flex for obstructive SFA disease | At 12 months post-index procedure
  Rate of stent fractures at 12 months post-index procedure
Rate of stent fractures at 12 months by type post-index procedure in patients treated with SMART Flex for obstructive PPA disease | At 12 months post-index procedure
  Rate of stent fractures at 12 months post-index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nusrath Sultana, Study Director — Cordis US Corp.
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided